CLINICAL TRIAL: NCT00117975
Title: A Phase II Trial of Extended Induction Galiximab (Anti-CD80 Monoclonal Antibody) (IND #12373) Plus Rituximab in Previously Untreated Follicular Non-Hodgkin Lymphoma (NHL)
Brief Title: Rituximab and Galiximab in Treating Patients With Stage II, Stage III, or Stage IV Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-50402; U10CA031946 (NIH); CDR0000433340 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2005-07-08; First posted 2005-07-11 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Lymphoma
Keywords: contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular | interventions — galiximab; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: galiximab — given IV
Biological: rituximab — Given IV

SUMMARY:
RATIONALE: Monoclonal antibodies, such as rituximab and galiximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving more than one monoclonal antibody may be a better way to block cancer growth.

PURPOSE: This phase II trial is studying how well giving rituximab together with galiximab works in treating patients with stage II, stage III, or stage IV non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the overall and complete response rate in patients with previously untreated CD20-positive bulky stage II or stage III or IV follicular non-Hodgkin's lymphoma treated with rituximab and galiximab.
* Determine the time to disease progression in patients treated with this regimen.

Secondary

* Determine the toxicity profile of this regimen in these patients.
* Correlate Fc receptor polymorphism profiling with response in patients treated with this regimen.

OUTLINE: This is a multicenter study.

* Induction therapy (month 1): Patients receive rituximab IV on days 1, 8, 15, and 22 and galiximab IV over 1 hour on day 3, 8, 15, and 22.
* Extended induction therapy (months 3, 5, 7, and 9): Beginning in month 3, patients receive rituximab and galiximab as above on day 1. Treatment repeats every 56 days for 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 4 months for up to 10 years.

PROJECTED ACCRUAL: A total of 51 patients will be accrued for this study within 18 months.

ELIGIBILITY:
1. Documentation of Disease

   1.1 Previously untreated, histologically confirmed follicular lymphoma, WHO classification, grade 1, 2, or 3a (> 15 centroblasts per high power field with centrocytes present) which is stage III, IV, or bulky (i.e., single mass ≥ 7 cm in any unidimensional measurement) stage II.

   1.1.1 Bone marrow biopsies as the sole means of diagnosis are not acceptable, but they may be submitted in conjunction with nodal biopsies. Fine needle aspirates are not acceptable.

   1.1.2 Failure to submit pathology specimens within 60 days of patient registration will result in the patient being declared ineligible.

   1.2 Institutional flow cytometry or immunohistochemistry must confirm CD20 antigen expression.

   1.3 Patients classified as high risk according to the Follicular Lymphoma International Prognostic Index (FLIPI) should be considered for CALGB 50102/SWOG S0016 (A Phase III Trial of CHOP vs CHOP + Rituximab vs CHOP + Iodine-131-Labeled Monoclonal Anti-B1 Antibody [Tositumomab] For Treatment of Newly Diagnosed Follicular Non-Hodgkin's Lymphomas).
2. Prior Treatment

   2.1 No prior therapy for non-Hodgkin lymphoma including chemotherapy, radiation or immunotherapy (e.g., monoclonal antibody-based therapy)

   2.2 No corticosteroids within two weeks prior to study, except for maintenance therapy for a non-malignant disease
3. Age - Patients must be ≥ 18 years of age
4. ECOG Performance Status - Patients must have ECOG Performance Status 0-2.
5. Measurable Disease - Measurable disease must be present either on physical examination or imaging studies.

   5.1 Non-measurable disease alone is not acceptable.

   5.2 Any tumor mass > 1 cm is acceptable.

   5.3 Lesions that are considered non-measurable include the following:
   * Bone lesions (lesions if present should be noted)
   * Ascites
   * Pleural/pericardial effusion
   * Lymphangitis cutis/pulmonis
   * Bone marrow (involvement by non-Hodgkin lymphoma should be noted).
6. CNS Involvement - Patients must have no known CNS involvement by lymphoma.
7. HIV Infection - Patients must have no known HIV infection.

   7.1 Patients with a history of intravenous drug abuse or any behavior associated with an increased risk of HIV infection should be tested for exposure to the HIV virus.

   7.2 Patients who test positive or who are known to be infected are not eligible due to an increased risk of infection with this regimen. An HIV test is not required for entry on this protocol, but is required if the patient is perceived to be at risk.
8. Human Anti-Chimeric Antibody - Patients must have no known baseline human anti-chimeric antibody (HACA) positivity.
9. Pregnancy and Nursing Status - Patients must be non-pregnant and non-nursing.

   9.1 Due to the unknown teratogenic potential of galiximab, pregnant or nursing patients may not be enrolled.

   9.2 Women and men of reproductive potential should agree to use an effective means of birth control throughout their participation in this study.

   9.3 Appropriate methods of birth control include oral contraceptives, implantable hormonal contraceptives, or double barrier method (diaphragm plus condom).
10. Second Malignancy - Patients with a "currently active" second malignancy, other than non-melanoma skin cancers are not eligible.

    10.1 This includes Waldenstrom's Macroglobulinemia, since such patients have experienced transient increases in IgM following initiation of rituximab, with the potential for hyperviscosity syndrome requiring plasmapheresis.

    10.2 Patients are not considered to have a "currently active" malignancy if they have completed anti-cancer therapy, and are considered by their physician to be at less than 30% risk of relapse.
11. Required Initial Laboratory Values:

    * ANC ≥ 1000/µL
    * Platelet Count ≥ 50,000/µL
    * Creatinine ≤ 2 x ULN Unless attributable to lymphoma
    * Total Bilirubin ≤ 2 x ULN*† Unless attributable to Gilbert's disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2005-06; Primary Completion 2007-06 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Overall response | 12 months
  complete and partial response will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Myron S. Czuczman, MD, Study Chair — Roswell Park Cancer Institute
Locations (68):
- United States (68):
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Michael & Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Iowa Blood and Cancer Care, Cedar Rapids, Iowa
  - St. Luke's Hospital, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - CancerCare of Maine at Eastern Maine Medial Center, Bangor, Maine
  - UMASS Memorial Cancer Center - University Campus, Worcester, Massachusetts
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Capital Region Cancer Center, Jefferson City, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - New Hampshire Oncology-Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Kingsbury Center for Cancer Care at Cheshire Medical Center, Keene, New Hampshire
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Elliot Regional Cancer Center, Manchester, New Hampshire
  - Frisbie Memorial Hospital, Rochester, New Hampshire
  - Roswell Park Cancer Institute, Buffalo, New York
  - Charles R. Wood Cancer Center at Glens Falls Hospital, Glens Falls, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - CCOP - Hematology-Oncology Associates of Central New York, Syracuse, New York
  - Community General Hospital of Greater Syracuse, Syracuse, New York
  - CaroMont Cancer Center at Gaston Memorial Hospital, Gastonia, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - Lenoir Memorial Cancer Center, Kinston, North Carolina
  - Wilson Medical Center, Wilson, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University, Columbus, Ohio
  - Western Pennsylvania Cancer Institute at Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - McLeod Regional Medical Center, Florence, South Carolina
  - Bon Secours St. Francis Health System, Greenville, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Mountainview Medical, Berlin Corners, Vermont
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Danville Regional Medical Center, Danville, Virginia
  - Ravenel Oncology Center at Memorial Hospital of Martinsville and Henry County, Martinsville, Virginia
  - St. Mary's Regional Cancer Center at St. Mary's Medical Center, Huntington, West Virginia

REFERENCES:
- [Result] Czuczman MS, Leonard JP, Johnson JL, et al.: FLIPI score is applicable and predictive of response to upfront immunotherapy in CALGB 50402: phase II trial of extended induction galiximab ([G] anti-CD80 monoclonal antibody) plus rituximab [R]. [Abstract] Blood 112 (11): A-1003, 2008.
- [Derived] Lansigan F, Barak I, Pitcher B, Jung SH, Cheson BD, Czuczman M, Martin P, Hsi E, Schoder H, Smith S, Bartlett NL, Leonard JP, Blum KA. The prognostic significance of PFS24 in follicular lymphoma following firstline immunotherapy: A combined analysis of 3 CALGB trials. Cancer Med. 2019 Jan;8(1):165-173. doi: 10.1002/cam4.1918. Epub 2018 Dec 21. PMID 30575311